CLINICAL TRIAL: NCT06757816
Title: Outcome of Accessory Rods and Ilic Fixation for Distal Augmentation of S1 Fixation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebram Eissa Moussa, principal investigator and resident orthopedic surgeon at Assiut university hospitals, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: accessory rods and iliac screw
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Lumbosacral
Keywords: accessory; fixation; rod; iliac; screws; L5; S1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A case series of patients who underwent extension of fixation for L5 S1 fusion (Other)
  Interventions: Procedure: accessory rod and iliac fixation for distal augmentation for S1 fixation.

INTERVENTIONS:
Procedure: accessory rod and iliac fixation for distal augmentation for S1 fixation. — patients who were admitted to the spine unit and needed extension of fixation for L5 S1 fusion due to failed previous surgery, instability, or degenerative changes ,infection, tumors and pseudoarthrosis.

SUMMARY:
To assess radiological and clinical outcome of use of accessory rod and iliac fixation for distal augmentation of L1 fixation

DETAILED DESCRIPTION:
Lumbar fusion is a surgical procedure that can be utilized to treat a variety of painful and degenerative conditions in the lower back. The most common conditions that indicate the need for an L5 S1 fusion include low back disc degeneration (also known as spondylolisthesis), spinal fractures, recurrent disc herniation, scoliosis, lumbar canal stenosis, and instability resulting from failed spine surgery . The success rate of lumbo sacral fusion surgery is influenced by many factors. These include non-union, hardware breakage or loosening, discitis, osteoporosis, tumors, and pseudoarthrosis . Lumbosacral pseudarthrosis is one of the most common complications in L5 S1 fusion surgery. It is a strong indication for revision surgery if severe symptoms persist. The rate of pseudarthrosis increases based on several parameters, including the number of levels fused, the type of fusion, and medical risk factors for pseudarthrosis .

There are various methods of revision. One such method involves the use of iliac screws in addition to lumbo sacral interbody fusion. This approach improves the outcomes of revision fusion surgery but still carries the risk of rod breakage . S2 alar-iliac (S2AI) screws have been described as another method, but they have some disadvantages like rod breakage, screw misplacement, breach of cortical bone, and injury to neurovascular structures. These structures include superior gluteal vessels, external iliac vessels, pudendal vessels, superior gluteal nerves, sciatic nerve, and sympathetic chain ganglia . Our theory proposes the use of an accessory rod, which offers the advantage of dual rod fixation with a low incidence of rod breakage. We also suggest the free-handed placement of the iliac screw in the iliac bone, which plays a significant role in improving the integrity of the fixation and simplifies the application process.

Multiple-rod constructs could prevent rod breakage and pseudarthrosis while also lowering the revision rate. As a result, they could lead to a better clinical outcome than the 2-rod construct. This approach is based on the principle that increasing the number of rods in the construct can distribute the load more evenly, reducing the risk of rod breakage and pseudarthrosis. This, in turn, could lead to a lower revision rate and better clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* The study will include all patients who were admitted to the spine unit and needed extension of fixation for L5 S1 fusion due to failed previous surgery, instability, or degenerative changes ,infection, tumors and pseudoarthrosis.

Exclusion Criteria:

* The study excludes patients who are less than 18 years and more than 90 years

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Outcome of accessory rod and iliac fixation for distal augmentation of S1 fixation | 3 months post-operative: Initial assessment of the union. 1 year post-operative: Follow-up to confirm sustained union and assess long-term outcomes.
  Union of L5 S1: This outcome is assessed by the presence of bridging bone across the fusion site, evaluated through X-ray imaging.

SECONDARY OUTCOMES:
Pain Relief | Preoperative: VAS scores will be recorded before the surgery. Immediate Postoperative: VAS scores will be recorded immediately after the surgery. 3 Months Postoperative: VAS scores will be recorded to evaluate changes in pain intensity.
  his will be assessed by comparing the preoperative and postoperative Visual Analogue Scale (VAS) scores of each patient. The VAS scores will be recorded before the surgery, immediately after the surgery, and at 3 months post-operative to evaluate changes in pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] Thomson S. Failed back surgery syndrome - definition, epidemiology and demographics. Br J Pain. 2013 Feb;7(1):56-9. doi: 10.1177/2049463713479096. PMID 26516498
- [Background] Herkowitz HN, Kurz LT. Degenerative lumbar spondylolisthesis with spinal stenosis. A prospective study comparing decompression with decompression and intertransverse process arthrodesis. J Bone Joint Surg Am. 1991 Jul;73(6):802-8. PMID 2071615
- [Background] Chakravarty A. A survey of attitude of frontline clinicians and nurses towards adverse events. Med J Armed Forces India. 2013 Oct;69(4):335-40. doi: 10.1016/j.mjafi.2013.01.009. Epub 2013 May 9. PMID 24600139
- [Background] Gill K, Blumenthal SL. Functional results after anterior lumbar fusion at L5-S1 in patients with normal and abnormal MRI scans. Spine (Phila Pa 1976). 1992 Aug;17(8):940-2. doi: 10.1097/00007632-199208000-00012. PMID 1387975